CLINICAL TRIAL: NCT06794970
Title: Tissue Study on the Chronic Active Humoral Rejection (cAMR) Population of Kidney Transplantation
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CARO Study
Record Dates: First submitted 2024-12-30; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is tissue-based, retrospective and prospective, single-centre, non-sponsored.

Primary objective: To examine patient and organ survival and eGFR variation in kidney transplant patients diagnosed histologically with cAMR.

DETAILED DESCRIPTION:
At the kidney transplant follow-up clinic of the UO Nephrology, Dialysis and Transplantation Unit of the IRCCS AOUBO Policlinico di Sant'Orsola, directed by Prof. G. La Manna, all patients with a diagnosis of cAMR made since 01/01/2018 and patients with a new diagnosis of cAMR made after the approval of this protocol by the Ethics Committee will be enrolled.

The study will last 5 years and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Kidney transplant recipients
* eGFR>15 ml/min/1.73 sq m at the time of diagnosis of cAMR
* cAMR diagnosis defined on the basis of the 2018 Banff Classification (17), made after 1/1/2018.
* Obtaining Informed Consent to Participation.

Exclusion Criteria:

* Combined transplant patients (heart-kidney, liver-kidney or kidney-pancreas)
* Histological evidence of concomitant disease (e.g. recurrence of original nephropathy or diagnosis of 'de novo' nephropathy, acute cellular rejection, polyomavirus BK nephropathy, other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the number of patients attending the Kidney Transplant Follow-up Outpatient Clinic of the Unit of Nephrology, Dialysis and Transplantation Prof. La Manna of the Policlinico di S. Orsola, about 50 patients will be enrolled, of whom about 25 have already been diagnosed and are undergoing treatment and about 25 new diagnoses are expected during the enrolment period in the prospective-only component.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Kidney survival post tranplant | 1 year, 2 years
  Patient and organ survival status
Change in eGFR | 1 year, 2 years
  The change in eGFR will be assessed by the linear slope of eGFR (least square method) in patients who have at least 3 serum creatinine assessments. In addition to the mean annual change in eGFR from the baseline visit, it will be assessed how many patients achieved a reduction in eGFR of 40% and 50% (percentage change) between the baseline visit and the 1- and 2-year follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Sant'Orsola University Hospital - Nephrology, Dialysis and Transplant Unit, Bologna, BO, Italy